CLINICAL TRIAL: NCT00379912
Title: Phase II Randomized Trial With A Modified Dose & Schedule of Subcutaneously Administered Azacitidine & Erythropoietin v Azacitidine Alone in Patients With Low-Risk Myelodysplastic Syndromes (Less Than 11% Marrow & Peripheral Blood Blasts)
Brief Title: Azacitidine and Erythropoietin Versus Azacitidine Alone for Patients With Low-Risk Myelodysplastic Syndromes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient response rate
Sponsor: Larry Cripe, MD (Other)
Collaborators: Celgene Corporation (Industry); Ortho Biotech Clinical Affairs, L.L.C. (Industry); Walther Cancer Institute (Other)
Responsible Party: Sponsor-Investigator, Larry Cripe, MD, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOG MDS04-85
Record Dates: First submitted 2006-09-21; First posted 2006-09-25 (Estimated); Results first posted 2017-05-31 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-01

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Azacitidine; Erythropoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Investigational Arm A (Experimental): Azacitidine + Erythropoietin
  Interventions: Drug: Azacitidine; Drug: Erythropoietin
- Investigational Arm B (Experimental): Azacitidine
  Interventions: Drug: Azacitidine (Monotherapy)

INTERVENTIONS:
Drug: Azacitidine — Azacitidine 50 mg/m2 subcutaneously qod for two consecutive weeks every four weeks.
  Other Names: Vidaza
  Arms: Investigational Arm A
Drug: Erythropoietin — Erythropoietin 60,000IU subcutaneous injection weekly while on protocol therapy
  Other Names: EPO
  Arms: Investigational Arm A
Drug: Azacitidine (Monotherapy) — Azacitidine 50 mg/m2 subcutaneously qod for two consecutive weeks every four weeks.
  Other Names: Vidaza
  Arms: Investigational Arm B

SUMMARY:
This trial is designed to explore a modified dose and schedule of azacitidine in order to more effectively address the needs of patients with low-risk myelodysplastic syndromes (MDS), i.e., to alter the natural history of the disease without excessive toxicity or burden. The administration of erythropoietin is designed to influence the differentiation of primitive hematopoietic cells in which azacitidine has reversed the abnormal phenotype to red blood cells for patients in whom inadequate production of red blood cells is the major clinical issue.

DETAILED DESCRIPTION:
OUTLINE: This is an open label, multi-center, randomized study.

Eligible patients will be randomized to one of two treatment arms:

Arm A (Azacitidine + Erythropoietin)

* Azacitidine Treatment 50 mg/m2 subcutaneously every other day (three times a week) for two consecutive weeks every four weeks. A cycle of therapy is defined as two consecutive weeks of subcutaneous azacitidine administered every other day three times a week (e.g. Monday - Wednesday - Friday) and the time to resolution of any treatment associated toxicity.
* Erythropoietin Treatment Patients who are randomized to Arm A will receive a dose of 60,000IU as a single subcutaneous injection weekly without interruption while enrolled on protocol therapy. The dose should be administered to coincide with the first day of each cycle.
* Protocol therapy may be administered for up to six cycles of therapy.

Arm B (Azacitidine Alone)

* Azacitidine Treatment 50 mg/m2 subcutaneously every other day (three times a week) for two consecutive weeks every four weeks. A cycle of therapy is defined as two consecutive weeks of subcutaneous azacitidine administered every other day three times a week (e.g. Monday - Wednesday - Friday) and the time to resolution of any treatment associated toxicity.
* Protocol therapy may be administered for up to six cycles of therapy.

ECOG performance status 0 to 2

Hematopoietic:

To be eligible for randomization, subjects must have documentation of at least 1 of the following:

* A transfusion dependent anemia (defined by a history of two or more episodes of transfusion within a period of 8 weeks).
* An untransfused hemoglobin < 10 gm/dl measured on at least two occasions more than 7 days apart in the month prior to randomization.

Patients must also meet 1 of the following criteria:

* Has not received prior erythropoietin and has a serum erythropoietin level > 200 IU/L within 14 days of randomization.
* Has received prior erythropoietin without clinical benefit in the judgment of the treating physician.
* Adequate iron status defined as serum ferritin > 20 ng/ml and transferrin saturation of > 30% within 90 days prior to randomization.
* Symptoms attributed to the anemia with hemoglobin < 11 g/dL.
* Folate and Vitamin B12 levels within normal limits within 90 days prior to randomization.

Hepatic:

* SGOT (ALT) level < 2 x ULN within 14 days prior to randomization.
* SGPT (AST) level < 2 x ULN within 14 days prior to randomization.
* Serum total bilirubin level < 2 x ULN within 14 days prior to randomization.

Renal:

* Serum creatine < 1.5 x the upper limit of normal (ULN) within 14 days prior to randomization.

Cardiovascular:

* No uncontrolled hypertension (defined as a systolic pressure > 160 mmHg and/or a diastolic pressure > 110 mmHg).
* No history of (within 12 months) deep venous thrombosis (DVT), pulmonary embolism (PE), or other venous thrombosis. Prior superficial thrombophlebitis is not an exclusion criterion.
* No history of (within 6 months) cerebrovascular accident ([CVA] includes ischemic, embolic, and hemorrhagic), transient ischemic attack (TIA), myocardial ischemia (includes Unstable Angina, Q wave Myocardial Infarction [QwMI], and non-Q wave Myocardial Infarction [NQMI]), or other arterial thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* A bone marrow (BM) aspirate and biopsy that demonstrates MDS with less than 11% blasts.
* Conventional metaphase cytogenetics done within 90 days prior to registration for screening.
* Central pathology review, correlative submission and confirmation of diagnosis is required prior to initiation of therapy (see Study Procedure Manual for details of submission). The FAB and WHO classification of MDS and the IPSS score will be determined at time of central pathology review.
* Correlative marrow aspirate obtained.

To be eligible for randomization, subjects must have documentation of at least 1 of the following:

* A transfusion dependent anemia (defined by a history of two or more episodes of transfusion within a period of 8 weeks).
* An untransfused hemoglobin < 10 gm/dl measured on at least two occasions more than 7 days apart in the month prior to randomization.

Patients must also meet 1 of the following criteria:

* Has not received prior erythropoietin and has a serum erythropoietin level > 200 IU/L within 14 days of randomization.
* Has received prior erythropoietin without clinical benefit in the judgment of the treating physician.
* Adequate iron status defined as serum ferritin > 20 ng/ml and transferrin saturation of > 30% within 90 days prior to randomization.
* Symptoms attributed to the anemia with hemoglobin < 11 g/dL.
* Folate and Vitamin B12 levels within normal limits within 90 days prior to randomization.
* Life expectancy > 6 months as judged by the treating investigator.

Exclusion Criteria:

* No known history of intolerance to erythropoietic agents.
* No prior intensive cytotoxic chemotherapy for a myeloid malignancy including MDS.
* Patients with a history of a non-myeloid malignancy with secondary MDS are eligible for study enrollment provided, in the opinion of the treating investigator and the study chair, the anticipated behavior of the non-myeloid malignancy will not interfere with study participation and evaluation of outcome.
* No known or suspected hypersensitivity to azacitidine or mannitol.
* No hepatic tumors.
* No uncontrolled hypertension (defined as a systolic pressure > 160 mmHg and/or a diastolic pressure > 110 mmHg).
* No known hypersensitivity to mammalian cell-derived products or human albumin.
* No history of (within 12 months) deep venous thrombosis (DVT), pulmonary embolism (PE), or other venous thrombosis. Prior superficial thrombophlebitis is not an exclusion criterion.
* No history of (within 6 months) cerebrovascular accident ([CVA] includes ischemic, embolic and hemorrhagic), transient ischemic attack (TIA), myocardial ischemia (includes Unstable Angina, Q wave Myocardial Infarction [QwMI] and non-Q wave Myocardial Infarction [NQMI], or other arterial thrombosis.
* Females of childbearing potential and males must be willing to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) while on treatment and for a 4-week period thereafter.
* Females with childbearing potential must have a negative pregnancy test within 7 days prior to being randomized. Patients are considered not of child bearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry Cripe, M.D., Study Chair — Hoosier Oncology Group, LLC
Locations (9):
- United States (9):
  - Medical & Surgical Specialists, LLC, Galesburg, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Quality Cancer Center (MCGOP), Indianapolis, Indiana
  - Arnett Cancer Care, Lafayette, Indiana
  - Horizon Oncology Center, Lafayette, Indiana
  - Medical Consultants, P.C., Muncie, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Center for Hematology-Oncology of S Michigan, Jackson, Michigan
  - Methodist Cancer Center, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sayar H, Chan RJ, Orschell CM, Chan EM, Yu Z, Hood D, Plett A, Yang Z, Hui CL, Nabinger SC, Kohlbacher KJ, West ES, Walter A, Sampson C, Wu J, Cripe LD. Thrice weekly azacitidine does not improve hematological responses in lower-risk myelodysplastic syndromes: a study of the Hoosier Oncology Group. Leuk Res. 2011 Aug;35(8):1108-10. doi: 10.1016/j.leukres.2011.02.025. Epub 2011 Mar 21. PMID 21420732
- See also: Hoosier Oncology Group Home Page — http://www.hoosieroncologygroup.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A Azacitidine + Erythropoietin: Azacitidine + Erythropoietin
  Azacitidine: Azacitidine 50 mg/m2 subcutaneously qod for two consecutive weeks every four weeks.
  Erythropoietin: Erythropoietin 60,000IU subcutaneous injection weekly while on protocol therapy
- Arm B Azacitidine: Azacitidine
  Azacitidine (Monotherapy): Azacitidine 50 mg/m2 subcutaneously qod for two consecutive weeks every four weeks.
Period: Overall Study
Arm/Group | Arm A Azacitidine + Erythropoietin | Arm B Azacitidine
Started | 7 | 8
Completed | 6 | 8
Not Completed | 1 | 0
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A Azacitidine + Erythropoietin | Arm B Azacitidine | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Continuous [Median (Full Range); unit: years] | 69 [63 to 85] | 67.50 [59 to 83] | 69 [59 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 6 | 7 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 8 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 8 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Overall Response After Cycle 3
Description: Overall response for participants who have completed at least three cycles of protocol-specified therapy according to the International Working Group to Standardize Response Criteria for Myelodysplastic Syndromes criteria for Erythroid Response (HI-E) Major response: For patients with pretreatment hemoglobin less than 11 g/dL, greater than 2 g/dL increase in hemoglobin; for RBC transfusion-dependent patients, transfusion independence.
  Minor response: For patients with pretreatment hemoglobin less than 11 g/dL, 1 to 2 g/dL increase in hemoglobin; for RBC transfusion-dependent patients, 50% decrease in transfusion requirements.
Time Frame: 3 months
Population: Participants completing at least three cycles at the time of analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants responding
Arm/Group | Arm A Azacitidine + Erythropoietin | Arm B Azacitidine
Number analyzed (Participants) | 6 | 6
percentage of participants responding | 50 [15.3 to 84.7] | 33.3 [6.3 to 72.9]

2. Primary Outcome: Overall Response Rate After Six Cycles
Description: Overall response rate for participants who have completed at least six cycles of protocol-specified therapy according to the International Working Group to Standardize Response Criteria for Myelodysplastic Syndromes criteria for Erythroid Response (HI-E) Major response: For patients with pretreatment hemoglobin less than 11 g/dL, greater than 2 g/dL increase in hemoglobin; for RBC transfusion-dependent patients, transfusion independence.
  Minor response: For patients with pretreatment hemoglobin less than 11 g/dL, 1 to 2 g/dL increase in hemoglobin; for RBC transfusion-dependent patients, 50% decrease in transfusion requirements.
Time Frame: 6 months
Population: Participants completing at least six cycles at the time of analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants responding
Arm/Group | Arm B Azacitidine | Arm A Azacitidine + Erythropoietin
Number analyzed (Participants) | 6 | 6
percentage of participants responding | 33.3 [6.3 to 72.9] | 33.3 [6.3 to 72.9]

3. Secondary Outcome: Safety Profile of the Modified Dose/Schedule of Azacitidine and Erythropoietin or a Modified Dose of Azacitidine Alone
Description: Full adverse event information is submitted in the record below. A summary of the Significant Toxicities Rate (clinically significant myelosuppression (CTCAE Grade 3 or 4 neutropenia or thrombocytopenia)) over all patients receiving at least 1 dose of study medication at the time of interim analysis is reported in this outcome measure.
Time Frame: 24 months
Population: All patients receiving at least 1 dose of study medication at the time of interim analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A Azacitidine + Erythropoietin | Arm B Azacitidine
Number analyzed (Participants) | 6 | 6
percentage of participants | 66.7 [27.1 to 93.7] | 66.4 [27.1 to 93.7]

4. Secondary Outcome: Duration of Significant Responses
Description: Data for this outcome measure was not collected or analyzed due to the termination of the study.
Time Frame: 24 months
Arm/Group | Arm A Azacitidine + Erythropoietin | Arm B Azacitidine
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Quality of Life
Description: Data for this outcome measure was not collected or analyzed due to the termination of the study
Time Frame: 24 months
Arm/Group | Investigational Arm A | Investigational Arm B
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Analysis of CD34, CD71, CD36 Cells in Aspirated Bone Marrow for Both Responders and Non-responders at Baseline and After Three and Six Cycles
Time Frame: 6 months
Population: Analysis of CD34, CD71, and CD36 cells was undertaken irrespective of arm assignment.
Measure: Mean (Standard Error); unit: cells of BM (10e^6/ML)
Groups:
- Responders: Responders
- Non-Responders: Non-Responders
Arm/Group | Responders | Non-Responders
Number analyzed (Participants) | 6 | 8
cells of BM (10e^6/ML)
  CD34 Baseline | .86 (.56) | .49 (.38)
  CD34 After Three Cycles | .93 (.78) | .58 (.28)
  CD34 After Six Cycles | 1.15 (.59) | .52 (.39)
  CD71 at Baseline | 18.32 (5.30) | 7.23 (3.32)
  CD71 After Three Cycles | 27.31 (14.33) | 10.13 (5.85)
  CD71 After Six Cycles | 35.45 (16.50) | 9.69 (7.36)
  CD36 at Baseline | 11.69 (2.76) | 5.12 (1.94)
  CD36 after Three Cycles | 14.33 (6.64) | 6.08 (4.27)
  CD36 after Six Cycles | 21.35 (9.23) | 3.57 (1.01)

7. Secondary Outcome: Percent Apoptosis in 34+36+71+ Cells at Baseline, Three Cycles and Six Cycles
Time Frame: Six months
Population: Analysis of percent apoptosis was undertaken irrespective of arm assignment and categorized between responsers and non-responders
Measure: Mean (Standard Error); unit: percentage of cells
Arm/Group | Responders | Non-Responders
Number analyzed (Participants) | 6 | 8
percentage of cells
  % apoptosis at baseline | 17.04 (6.04) | 31.19 (12.03)
  % apoptosis after three cycles | 24.70 (9.01) | 63.43 (7.72)
  % apoptosis after six cycles | 42.58 (11.41) | 38.10 (4.84)

8. Secondary Outcome: BclXL Expression
Time Frame: Six months
Population: Analysis of BclXL expression was undertaken irrespective of arm assignment and categorized between responsers and non-responders
Measure: Mean (Standard Error); unit: percentage L27 mRNA
Arm/Group | Responders | Non-Responders
Number analyzed (Participants) | 6 | 8
percentage L27 mRNA
  BclXL Expression at baseline | 1.0 (0.00) | 1.00 (0)
  BclXL Expression after three cycles | 1.50 (0.32) | .77 (.15)
  BclXL Expression after six cycles | 3.89 (.99) | 1.21 (.37)

ADVERSE EVENTS:
Time Frame: The duration of study participation, up to two years
Arm/Group | Arm A Azacitidine + Erythropoietin | Arm B Azacitidine
Serious Adverse Events (participants affected / at risk) | 4/7 | 2/8
Other Adverse Events (participants affected / at risk) | 7/7 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A Azacitidine + Erythropoietin (N=7) | Arm B Azacitidine (N=8)
ENTERITIS (INFLAMMATION OF THE SMALL BOWEL) (Gastrointestinal disorders) | 1 (1) | 0 (0)
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 0 (0) | 1 (1)
HEMORRHAGE, GI / UPPER GI NOS (Gastrointestinal disorders) | 0 (0) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / BLADDER (URINARY) (Infections and infestations) | 0 (0) | 1 (1)
PLEURAL EFFUSION (NON-MALIGNANT) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA / ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0)
TUMOR LYSIS SYNDROME (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A Azacitidine + Erythropoietin (N=7) | Arm B Azacitidine (N=8)
ALLERGIC RHINITIS (INCLUDING SNEEZING, NASAL STUFFINESS, POSTNASAL DRIP) (Immune system disorders) | 0 (0) | 2 (2)
ANOREXIA (Gastrointestinal disorders) | 1 (1) | 2 (2)
ARTHRITIS (NON-SEPTIC) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
AUDITORY/EAR (Ear and labyrinth disorders) | 1 (1) | 0 (0)
BRUISING (IN ABSENCE OF GRADE 3 OR 4 THROMBOCYTOPENIA) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
CARDIAC ARRHYTHMIA (Cardiac disorders) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 4 (5)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 1 (1) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (1) | 1 (1)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2)
EDEMA: LIMB (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
ESOPHAGITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 4 (10) | 2 (4)
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 0 (0) | 1 (2)
HAIR LOSS/ALOPECIA (SCALP OR BODY) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
HEMATOMA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
HEMOGLOBIN (Blood and lymphatic system disorders) | 4 (15) | 7 (19)
HEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 1 (1)
HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
HYPERTENSION (Cardiac disorders) | 0 (0) | 1 (1)
HYPOTENSION (Cardiac disorders) | 0 (0) | 1 (1)
INFECTION WITH GRADE 3 OR 4 NEUTROPHILS (ANC <1.0 X 10E9/L) / ABDOMEN NOS (Infections and infestations) | 1 (1) | 0 (0)
INFECTION WITH GRADE 3 OR 4 NEUTROPHILS (ANC <1.0 X 10E9/L) / MIDDLE EAR (OTITIS MEDIA) (Infections and infestations) | 0 (0) | 1 (1)
INFECTION WITH GRADE 3 OR 4 NEUTROPHILS (ANC <1.0 X 10E9/L) / URINARY TRACT NOS (Infections and infestations) | 0 (0) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / LUNG (PNEUMONIA) (Infections and infestations) | 0 (0) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / URINARY TRACT NOS (Infections and infestations) | 0 (0) | 1 (1)
INJECTION SITE REACTION/EXTRAVASATION CHANGES (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
INSOMNIA (General disorders) | 0 (0) | 1 (1)
IRON OVERLOAD (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
LEUKOCYTES (TOTAL WBC) (Blood and lymphatic system disorders) | 1 (5) | 0 (0)
MOOD ALTERATION / ANXIETY (Psychiatric disorders) | 0 (0) | 1 (1)
MUCOSITIS/STOMATITIS (FUNCTIONAL/SYMPTOMATIC) / ORAL CAVITY (Gastrointestinal disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1)
NEUTROPHILS/GRANULOCYTES (ANC/AGC) (Blood and lymphatic system disorders) | 5 (15) | 5 (15)
PAIN / ABDOMEN NOS (Gastrointestinal disorders) | 1 (3) | 1 (1)
PAIN / BONE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN / EXTREMITY-LIMB (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
PAIN / GALLBLADDER (Hepatobiliary disorders) | 1 (1) | 0 (0)
PAIN / MIDDLE EAR (Ear and labyrinth disorders) | 0 (0) | 1 (1)
PAIN / NECK (General disorders) | 1 (1) | 0 (0)
PAIN (General disorders) | 0 (0) | 1 (1)
PLATELETS (Blood and lymphatic system disorders) | 3 (12) | 4 (24)
RIGORS/CHILLS (General disorders) | 0 (0) | 1 (2)
SWEATING (DIAPHORESIS) (General disorders) | 1 (1) | 0 (0)
URIC ACID, SERUM-HIGH (HYPERURICEMIA) (Investigations) | 1 (2) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (1)
WEIGHT LOSS (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Results of interim analysis led to early closure of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No